CLINICAL TRIAL: NCT00197054
Title: A Phase IIb Randomized, Double-blind, Controlled Study of the Safety, Immunogenicity and Proof-of-concept of RTS,S/AS02A, and RTS,S/AS01B, Two Candidate Malaria Vaccines in Malaria-experienced Adults Living in Western Kenya.
Brief Title: Safety, Immunogenicity of RTS,S/AS02A, and RTS,S/AS01B Malaria Vaccines in Malaria-experienced Adults.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: GlaxoSmithKline (Industry); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: A-12227; IND 11220 (Other: FDA)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2020-12-11 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Plasmodium Falciparum
MeSH Terms: conditions — Malaria, Falciparum | interventions — RTS,S-AS01B vaccine; RTS,S-AS02A vaccine; Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VACC 1 (RTS, S/AS01B) (Experimental): RTS, S/AS01B: 0.5mL dose; 50ug RTS, S antigen, 50ug QS21 and liposomes in phosphate-buffered saline administered intramuscular deltoid of non-dominant arm at 0, 1 and 2 months.
  Interventions: Biological: RTS, S/AS01B
- VACC 2 (RTS, S/AS02A) (Experimental): RTS, S/AS02A: 0.5mL dose; 50ug RTS, S antigen, 50ug QS21 and proprietary oil-water emulsion in phosphate-buffered saline administered intramuscular deltoid of non-dominant arm at 0, 1 and 2 months.
  Interventions: Biological: RTS, S/AS02A
- Rabipur (Rabies) Vaccine (Active Comparator): Rabipur (Rabies) Vaccine: 1.0mL dose administered intramuscular deltoid of non-dominant arm at 0, 1 and 2 months.
  Interventions: Biological: Rabipur (Rabies) Vaccine

INTERVENTIONS:
Biological: RTS, S/AS01B — 0.5mL dose; 50ug RTS, S antigen, 50ug QS21 and liposomes in phosphate-buffered saline administered intramuscular deltoid of non-dominant arm at 0, 1 and 2 months.
  Arms: VACC 1 (RTS, S/AS01B)
Biological: RTS, S/AS02A — 0.5mL dose; 50ug RTS, S antigen, 50ug QS21 and proprietary oil-water emulsion in phosphate-buffered saline administered intramuscular deltoid of non-dominant arm at 0, 1 and 2 months.
  Arms: VACC 2 (RTS, S/AS02A)
Biological: Rabipur (Rabies) Vaccine — 1.0mL dose administered intramuscular deltoid of non-dominant arm at 0, 1 and 2 months
  Arms: Rabipur (Rabies) Vaccine

SUMMARY:
The candidate malaria vaccine RTS,S/AS02A developed by GSK Biologicals demonstrated 30% efficacy against clinical episodes of malaria and approximately 58% efficacy against severe malaria disease. As a potential improvement to RTS,S/AS02A, another candidate vaccine RTS,S/AS01B is being developed in parallel in collaboration with the Walter Reed Army Institute of Research (WRAIR). This study will be the first administration of the RTS,S/AS01B vaccine to the African adults to establish safety and immunogenicity in this population. Preliminary indication of vaccine efficacy with this adjuvant will be established by monitoring the time to the first infection with Plasmodium falciparum.

DETAILED DESCRIPTION:
The study comprises of 3 groups and the participating subjects will be randomly allocated to one of the three groups. The first group will receive RTS,S/AS01B, the second group will receive RTS,S/AS02A and the third group will receive rabies vaccine. Immunization will be given by IM injection on 0, 1, 2 month schedule. Infants will be followed up daily for 7 days for solicited symptoms and 30 days for unsolicited symptoms after each vaccine dose. Serious adverse events will be recorded throughout the study period. A week prior to Dose 3, subjects will be treated with a licenced anti-malarial drug. Starting from two weeks after Dose 3, the subjects will be monitored for a 14-week duration for detection of malaria infection.

ELIGIBILITY:
Inclusion criteria:

* Healthy male or female volunteers aged between 18 and 35 years at the time of first vaccination who have given written consent for their participation in the study were included
* If the volunteer is female, she must be of non-childbearing potential, i.e. either surgically sterilized or one year post-menopausal; or, if of childbearing potential, she must be abstinent or have used adequate contraceptive precautions for 30 days prior to vaccination, have a negative pregnancy test and must agree to continue such precautions for two months after completion of the vaccination series

Exclusion criteria:

* If a subject plans to take vaccine not foreseen by the study protocol within 30 days of the first dose of vaccine(s) with the exception of tetanus toxoid will be excluded
* Volunteers with any confirmed or suspected immunosuppressive or immunodeficient conditions
* Family history of congenital or hereditary immunodeficiency
* History of allergic reactions to previous immunizations
* HBsAg positive subjects
* History of splenectomy
* Pregnant or lactating females will be excluded from the study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 255 (Actual)
Dates: Start 2005-07 (Actual); Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- U.S. Army Research Unit-Kenya, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: Yes
GSK and WRAIR
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Polhemus ME, Remich SA, Ogutu BR, Waitumbi JN, Otieno L, Apollo S, Cummings JF, Kester KE, Ockenhouse CF, Stewart A, Ofori-Anyinam O, Ramboer I, Cahill CP, Lievens M, Dubois MC, Demoitie MA, Leach A, Cohen J, Ballou WR, Heppner DG Jr. Evaluation of RTS,S/AS02A and RTS,S/AS01B in adults in a high malaria transmission area. PLoS One. 2009 Jul 31;4(7):e6465. doi: 10.1371/journal.pone.0006465. PMID 19649245

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 255 subjects were enrolled and randomized 1:1:1 into each arm at Kombewa Clinic, US Army Medical Research Unit, Kisumu Kenya.
Period: Overall Study
Arm/Group | RTS, S/AS02A | RTS, S/AS01B | Rabipur (Rabies) Vaccine
Started | 85 | 85 | 85
Completed | 68 | 64 | 73
Not Completed | 17 | 21 | 12
Not completed — Withdrawal by Subject | 9 | 3 | 3
Not completed — Moved from area | 7 | 14 | 9
Not completed — Lost to Follow-up | 1 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RTS, S/AS02A | RTS, S/AS01B | Rabipur (Rabies) Vaccine | Total
Number analyzed (Participants) | 85 | 85 | 85 | 255
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.2 (5.16) | 24.9 (5.50) | 26.1 (5.10) | 25.4 (5.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 12 | 52
  Male | 66 | 64 | 73 | 203
Region of Enrollment [Number; unit: participants]
  Kenya | 85 | 85 | 85 | 255

OUTCOME MEASURES:

1. Primary Outcome: Safety: Proportion of Subjects With Grade 3 Solicited and Unsolicited General Reactions After Vaccination of RTS, S/AS02A and RTS, S/AS01B
Description: Proportion of subjects with grade 3 solicited and unsolicited general reactions after vaccination of RTS, S/AS02A and RTS, S/AS01B during a 7 day follow-up period (day of vaccination + 6 days).
Time Frame: 7 day follow-up (day of vaccination + 6 days)
Population: Rabipur was a comparator vaccine and not relevant to results of this primary outcome. Results for Rabipur were not presented in data table.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | RTS, S/AS02A | RTS, S/AS01B
Number analyzed (Participants) | 85 | 85
participants | 0 [0.0 to 4.2] | 1 [0.0 to 6.4]

2. Primary Outcome: Safety: Number of Administered Doses Eliciting Grade 3 Unsolicited Symptoms
Description: Grade 3 unsolicited symptoms reported following any number of administered doses
Time Frame: 6.5 months
Measure: Number (95% Confidence Interval); unit: administered doses
Units Other Than Participants: Doses
Arm/Group | RTS, S/AS01B | RTS, S/AS02A | Rabipur (Rabies) Vaccine
Number analyzed (Participants) | 85 | 85 | 85
Number analyzed (Doses) | 242 | 247 | 247
administered doses
  At least one symptom | 3 [0.3 to 3.6] | 0 [0.0 to 1.5] | 1 [0.0 to 2.2]
  Sinusitis | 1 [0.0 to 2.3] | 0 [0.0 to 1.5] | 0 [0.0 to 1.5]
  Headache | 1 [0.0 to 2.3] | 0 [0.0 to 1.5] | 1 [0.0 to 2.2]
  Cough | 1 [0.0 to 2.3] | 0 [0.0 to 1.5] | 0 [0.0 to 1.5]

3. Primary Outcome: Safety: Number of Doses Eliciting Solicited Local Symptoms Reported Over 7 Day Follow-up Period
Description: Incidence overall solicited general and local reactions over 7 day follow-up period after dose 1, 2 and 3 (Total Cohort)
Time Frame: 7 day follow-up period (day of vaccination + 6 days)
Population: number of administered doses
Measure: Number; unit: Doses
Units Other Than Participants: Doses
Arm/Group | RTS, S/AS01B | RTS, S/AS02A | Rabipur (Rabies) Vaccine
Number analyzed (Participants) | 85 | 85 | 85
Number analyzed (Doses) | 242 | 247 | 247
Doses
  Pain | 132 | 166 | 68
  Swelling | 12 | 22 | 2
  Fatigue | 43 | 33 | 35
  Fever (Axillary) | 21 | 14 | 12
  Gastrointestinal | 48 | 42 | 44
  Headache | 84 | 95 | 67
  Joint pain at other location | 27 | 22 | 22
  Muscle aches | 27 | 23 | 29

4. Secondary Outcome: Safety: Occurrence of SAEs
Description: Percentage of subjects experiencing SAEs classified by MedRA System Organ Class and Preferred Term (Month 6.5-12)
Time Frame: months 6.5 thru 12
Population: Number of subjects with at least one administered dose
Measure: Number (95% Confidence Interval); unit: % of subjects
Arm/Group | RTS, S/AS01B | RTS, S/AS02A | Rabipur (Rabies) Vaccine
Number analyzed (Participants) | 74 | 76 | 76
% of subjects
  Anaemia | 1.4 [0.0 to 7.3] | 0.0 [0.0 to 4.7] | 0.0 [0.0 to 4.7]
  Cardiac Failure | 0.0 [0.0 to 4.9] | 0.0 [0.0 to 4.7] | 1.3 [0.0 to 7.1]
  Pericardial Effusion | 0.0 [0.0 to 4.9] | 0.0 [0.0 to 4.7] | 1.3 [0.0 to 7.1]
  Cataract | 0.0 [0.0 to 4.9] | 0.0 [0.0 to 4.7] | 1.3 [0.0 to 7.1]
  Wound Necrosis | 1.4 [0.0 to 7.3] | 0.0 [0.0 to 4.7] | 0.0 [0.0 to 4.7]
  Abscess Limb | 0.0 [0.0 to 4.9] | 0.0 [0.0 to 4.7] | 1.3 [0.0 to 7.1]
  HIV Infection | 1.4 [0.0 to 7.3] | 0.0 [0.0 to 4.7] | 1.3 [0.0 to 7.1]
  Lobar Pneumonia | 1.4 [0.0 to 7.3] | 0.0 [0.0 to 4.7] | 0.0 [0.0 to 4.7]
  Malaria | 0.0 [0.0 to 4.9] | 1.3 [0.0 to 7.1] | 0.0 [0.0 to 4.7]
  Meningitis | 1.4 [0.0 to 7.3] | 0.0 [0.0 to 4.7] | 1.3 [0.0 to 7.1]
  Pneumonia | 1.4 [0.0 to 7.3] | 0.0 [0.0 to 4.7] | 0.0 [0.0 to 4.7]
  Pulmonary Tuberculosis | 0.0 [0.0 to 4.9] | 0.0 [0.0 to 4.7] | 1.3 [0.0 to 7.1]
  Trichomoniasis | 1.4 [0.0 to 7.3] | 0.0 [0.0 to 4.7] | 0.0 [0.0 to 4.7]
  Abortion | 1.4 [0.0 to 7.3] | 0.0 [0.0 to 4.7] | 0.0 [0.0 to 4.7]
  Haemoptysis | 2.4 [0.0 to 7.3] | 0.0 [0.0 to 4.7] | 0.0 [0.0 to 4.7]
  Pleural Effusion | 0.0 [0.0 to 4.9] | 0.0 [0.0 to 4.7] | 1.3 [0.0 to 7.1]

5. Secondary Outcome: Safety: Occurrence of SAEs
Description: Percentage of subjects reporting SAEs classified by MedDRA System Organ Class and Preferred Term (Month 0-12)
Time Frame: months 0 thru 12
Population: Number of subjects with at least one administered dose
Measure: Number (95% Confidence Interval); unit: % of subjects reporting symptom
Arm/Group | RTS, S/AS01B | RTS, S/AS02A | Rabipur (Rabies) Vaccine
Number analyzed (Participants) | 85 | 85 | 85
% of subjects reporting symptom
  Anaemia | 1.2 [0.0 to 6.4] | 0.0 [0.0 to 4.2] | 0.0 [0.0 to 4.2]
  Cardiac Failure | 0.0 [0.0 to 4.2] | 0.0 [0.0 to 4.2] | 1.2 [0.0 to 6.4]
  Pericardial Effusion | 0.0 [0.0 to 4.2] | 0.0 [0.0 to 4.2] | 1.2 [0.0 to 6.4]
  Cataract | 0.0 [0.0 to 4.2] | 0.0 [0.0 to 4.2] | 1.2 [0.0 to 6.4]
  Peptic Ulcer Haemorrhage | 1.2 [0.0 to 6.4] | 0.0 [0.0 to 4.2] | 0.0 [0.0 to 4.2]
  Wound Necrosis | 1.2 [0.0 to 6.4] | 0.0 [0.0 to 4.2] | 0.0 [0.0 to 4.2]
  Abscess Limb | 0.0 [0.0 to 4.2] | 0.0 [0.0 to 4.2] | 1.2 [0.0 to 6.4]
  Disseminated Tuberculosis | 1.2 [0.0 to 6.4] | 0.0 [0.0 to 4.2] | 0.0 [0.0 to 4.2]
  HIV Infection | 2.4 [0.3 to 8.2] | 0.0 [0.0 to 4.2] | 3.5 [0.7 to 10.0]
  Lobar Pneumonia | 1.2 [0.0 to 6.4] | 0.0 [0.0 to 4.2] | 0.0 [0.0 to 4.2]
  Malaria | 0.0 [0.0 to 4.2] | 1.2 [0.0 to 6.4] | 0.0 [0.0 to 4.2]
  Meningitis | 1.2 [0.0 to 6.4] | 0.0 [0.0 to 4.2] | 1.2 [0.0 to 6.4]
  Meningitis Cryptococcal | 0.0 [0.0 to 4.2] | 0.0 [0.0 to 4.2] | 1.2 [0.0 to 6.4]
  Pneumocystis Jiroveci Pheumonia | 1.2 [0.0 to 6.4] | 0.0 [0.0 to 4.2] | 0.0 [0.0 to 4.2]
  Pneumonia | 1.2 [0.0 to 6.4] | 0.0 [0.0 to 4.2] | 0.0 [0.0 to 4.2]
  Pulmonary Tuberculosis | 0.0 [0.0 to 4.2] | 0.0 [0.0 to 4.2] | 1.2 [0.0 to 6.4]
  Trichomoniasis | 1.2 [0.0 to 6.4] | 0.0 [0.0 to 4.2] | 0.0 [0.0 to 4.2]
  Osteoarthritis | 1.2 [0.0 to 6.4] | 0.0 [0.0 to 4.2] | 0.0 [0.0 to 4.2]
  Encephalitis | 1.2 [0.0 to 6.4] | 0.0 [0.0 to 4.2] | 0.0 [0.0 to 4.2]
  Abortion | 1.2 [0.0 to 6.4] | 0.0 [0.0 to 4.2] | 0.0 [0.0 to 4.2]
  Haemoptysis | 1.2 [0.0 to 6.4] | 0.0 [0.0 to 4.2] | 0.0 [0.0 to 4.2]
  Pleural Effusion | 0.0 [0.0 to 4.2] | 0.0 [0.0 to 4.2] | 1.2 [0.0 to 6.4]

6. Secondary Outcome: Occurrence of Hematology Parameters Below Normal Range
Description: Occurrence of hematology parameters below normal range (Total Cohort)
Time Frame: Days 0, 6, 66, and 90; Months 6 and 12
Measure: Count of Participants; unit: Participants
Arm/Group | RTS, S/AS01B | RTS, S/AS02A | Rabipur (Rabies) Vaccine
Number analyzed (Participants) | 85 | 85 | 85
Participants
  Hemoglobin: Day 0 | 0 | 0 | 0
  Hemoglobin: Day 6 | 4 | 1 | 1
  Hemoglobin: Day 66 | 2 | 1 | 2
  Hemoglobin: Day 90 | 2 | 0 | 2
  hemoglobin: Month 6 | 2 | 1 | 1
  Hemoglobin: Month 12 | 4 | 2 | 0
  WBC: Day 0 | 0 | 0 | 0
  WBC: Day 6 | 0 | 0 | 1
  WBC: Day 66 | 0 | 0 | 1
  WBC: Day 90 | 3 | 0 | 0
  WBC: Month 6 | 2 | 0 | 1
  WBC: Month 12 | 2 | 0 | 0
  Lymphocytes: Day 0 | 0 | 0 | 0
  Lymphocytes: Day 6 | 0 | 0 | 1
  Lymphocytes: Day 66 | 0 | 0 | 0
  Lymphocytes: Day 90 | 1 | 0 | 0
  Lymphocytes: Month 6 | 1 | 0 | 0
  Lymphocytes: Month 12 | 1 | 0 | 0

7. Secondary Outcome: Occurrence of Biochemistry Parameters Above Normal Ranges
Description: Occurrence of parameters of biochemical monitoring above normal ranges (Total Cohort)
Time Frame: Days 0, 6, and 90
Measure: Count of Participants; unit: Participants
Arm/Group | RTS, S/AS01B | RTS, S/AS02A | Rabipur (Rabies) Vaccine
Number analyzed (Participants) | 85 | 85 | 85
Participants
  Bilirubin: Day 0 | 10 | 9 | 11
  Bilirubin: Day 6 | 6 | 4 | 7
  Bilirubin: Day 90 | 3 | 3 | 6
  ALT: Day 0 | 0 | 0 | 0
  ALT: Day 6 | 1 | 6 | 0
  ALT: Day 90 | 0 | 1 | 3

8. Other Pre Specified Outcome: Seropositivity Rates for Anti-HBs Antibodies by Infection Status PRE
Description: Seropositivity rates and GMTs for Anti-HBs antibodies by infection status (Total Cohort) Seropositive >3.3 mlU/mL; Seroprotected >10 mIU/mL Infection defined as P. falciparum asexual parasitemia >0 PRE= Prevaccination
Time Frame: Prevaccination
Population: The Total Vaccinated Cohort includes all vaccinated subjects for whom data were available. For seropositivity rates by infection status arms have been combined.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- >=3.3 MIU/ML: Seropositive: >3.3 mlU/mL
- >=10 MIU/ML: Seroprotected: >10 mlU/mL
Arm/Group | >=3.3 MIU/ML | >=10 MIU/ML
Number analyzed (Participants) | 163 | 163
percentage of participants
  % of Non-infected: number analyzed (Participants) | 67 | 67
  % of Non-infected | 38.8 [27.1 to 51.5] | 37.3 [25.8 to 50.0]
  % of Infected: number analyzed (Participants) | 96 | 96
  % of Infected | 50.0 [39.6 to 60.4] | 44.8 [34.6 to 55.3]

9. Other Pre Specified Outcome: Seropositivity Rates for Anti-HBs Antibodies by Infection Status PIII(D90)
Description: Seropositivity rates and GMTs for Anti-HBs antibodies by infection status (Total Cohort) Seropositive >3.3 mlU/mL; Seroprotected: >10 mlU/mL Infection defined as P. falciparum asexual parasitemia >0 PIII(D90)= post dose 3 (day 90)
Time Frame: Day 90
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | >=3.3 MIU/ML | >=10 MIU/ML
Number analyzed (Participants) | 152 | 152
percentage of participants
  % of Non-infected: PIII(D90): number analyzed (Participants) | 57 | 57
  % of Non-infected: PIII(D90) | 96.5 [87.9 to 99.6] | 93.0 [83.0 to 98.1]
  % of Infected: PIII(D90): number analyzed (Participants) | 95 | 95
  % of Infected: PIII(D90) | 93.7 [86.8 to 97.6] | 91.6 [84.1 to 96.3]

10. Other Pre Specified Outcome: Seropositivity Rates for Anti-HBs Antibodies by Infection Status PIII(M12)
Description: Seropositivity rates and GMTs for Anti-HBs antibodies by infection status (Total Cohort) Seropositive >3.3 mlU/mL; Seroprotected: >10 mlU/mL Infection defined as P. falciparum asexual parasitemia >0 PIII(M12)= post dose 3 (month 12)
Time Frame: Month 12
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | >=3.3 MIU/ML | >=10 MIU/ML
Number analyzed (Participants) | 132 | 132
percentage of participants
  % of Non-infected: PIII(M12): number analyzed (Participants) | 47 | 47
  % of Non-infected: PIII(M12) | 97.9 [88.7 to 99.9] | 91.5 [79.6 to 97.6]
  % of Infected: PIII(M12): number analyzed (Participants) | 85 | 85
  % of Infected: PIII(M12) | 92.9 [85.3 to 97.4] | 90.6 [82.3 to 95.8]

11. Other Pre Specified Outcome: Seropositivity Rates for Anti-HBs Antibodies by Vaccine Group PRE
Description: Seropositivity rates for Anti-HBs antibodies by vaccine group (ATP Cohort for Immunogenicity).
  Seropositive >3.3 mlU/ML
  PRE=Prevaccination
Time Frame: Prevaccination
Population: Subject with available results
Measure: Count of Participants; unit: Participants
Arm/Group | RTS, S/AS01B | RTS, S/AS02A | Rabipur (Rabies) Vaccine
Number analyzed (Participants) | 73 | 70 | 68
Participants | 31 | 38 | 35

12. Other Pre Specified Outcome: Seropositivity Rates for Anti-HBs Antibodies by Vaccine Group PIII(D90)
Description: Seropositivity rates for Anti-HBs antibodies by vaccine group (ATP Cohort for Immunogenicity).
  Seropositive >3.3 mlU/ML
  PIII(D90)= post dose 3 (Day 90)
Time Frame: Day 90
Population: Subjects with available results
Measure: Count of Participants; unit: Participants
Arm/Group | RTS, S/AS01B | RTS, S/AS02A | Rabipur (Rabies) Vaccine
Number analyzed (Participants) | 72 | 72 | 65
Participants | 68 | 68 | 37

13. Other Pre Specified Outcome: Seropositivity Rates for Anti-HBs Antibodies by Vaccine Group PIII(M12)
Description: Seropositivity rates for Anti-HBs antibodies by vaccine group (ATP Cohort for Immunogenicity).
  Seropositive >3.3 mlU/ML
  PIII(M12)= post dose 3 (Month 12)
Time Frame: Month 12
Population: Subjects with available results
Measure: Count of Participants; unit: Participants
Arm/Group | RTS, S/AS01B | RTS, S/AS02A | Rabipur (Rabies) Vaccine
Number analyzed (Participants) | 61 | 62 | 66
Participants | 57 | 59 | 40

14. Other Pre Specified Outcome: Seroprotection Rates for Anti-HBs Antibodies by Vaccine Group PRE
Description: Seroprotection rates for Anti-HBs antibodies by vaccine group (ATP Cohort for Immunogenicity).
  Seroprotected >10 mlU/mL
  PRE=Prevaccination
Time Frame: Prevaccination
Population: Subjects with available results
Measure: Count of Participants; unit: Participants
Arm/Group | RTS, S/AS01B | RTS, S/AS02A | Rabipur (Rabies) Vaccine
Number analyzed (Participants) | 73 | 70 | 68
Participants | 29 | 34 | 33

15. Other Pre Specified Outcome: Seroprotection Rates for Anti-HBs Antibodies by Vaccine Group PIII (D90)
Description: Seroprotection rates for Anti-HBs antibodies by vaccine group (ATP Cohort for Immunogenicity).
  Seroprotected >10 mlU/mL
  PIII(D90)= post dose 3 (Day 90)
Time Frame: Day 90
Population: Subject with available results
Measure: Count of Participants; unit: Participants
Arm/Group | RTS, S/AS01B | RTS, S/AS02A | Rabipur (Rabies) Vaccine
Number analyzed (Participants) | 72 | 72 | 65
Participants | 65 | 67 | 33

16. Other Pre Specified Outcome: Seroprotection Rates for Anti-HBs Antibodies by Vaccine Group PIII (M12)
Description: Seroprotection rates for Anti-HBs antibodies by vaccine group (ATP Cohort for Immunogenicity).
  Seroprotected >10 mlU/mL
  PIII(M12)= post dose 3 (Month 12)
Time Frame: Month 12
Population: Subjects with available results
Measure: Count of Participants; unit: Participants
Arm/Group | RTS, S/AS01B | RTS, S/AS02A | Rabipur (Rabies) Vaccine
Number analyzed (Participants) | 61 | 62 | 66
Participants | 55 | 57 | 33

17. Other Pre Specified Outcome: Geometric Mean Antibody Titers (GMTs) for Anti-HBs Antibodies by Vaccine Group PRE
Description: Geometric mean antibody titers (GMTs) for Anti-HBs antibodies by vaccine group (According to protocol (ATP) Cohort for Immunogenicity)
  PRE=Prevaccination
Time Frame: Prevaccination
Population: Subjects with available results
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | RTS, S/AS01B | RTS, S/AS02A | Rabipur (Rabies) Vaccine
Number analyzed (Participants) | 73 | 70 | 68
titers | 11.1 [6.0 to 20.4] | 18.3 [9.4 to 35.3] | 23.6 [11.3 to 49.0]

18. Other Pre Specified Outcome: Geometric Mean Titers (GMTs) for Anti-HBs Antibodies by Vaccine Group PIII (D90)
Description: Geometric mean titers (GMTs) for Anti-HBs antibodies by vaccine group (According to protocol (ATP) Cohort for Immunogenicity)
  PIII(D90)= post dose 3 (Day 90)
Time Frame: Day 90
Population: Subjects with available results
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | RTS, S/AS01B | RTS, S/AS02A | Rabipur (Rabies) Vaccine
Number analyzed (Participants) | 72 | 72 | 65
titers | 1434.9 [743.0 to 2770.9] | 1714.3 [836.1 to 3515.0] | 31.7 [14.6 to 68.9]

19. Other Pre Specified Outcome: Geometric Mean Titers (GMTs) for Anti-HBs Antibodies by Vaccine Group PIII (M12)
Description: Geometric mean titers (GMTs) for Anti-HBs antibodies by vaccine group (According to protocol (ATP) Cohort for Immunogenicity)
  PIII(M12)= post dose 3 (Month 12)
Time Frame: Month 12
Population: Subjects with available results
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | RTS, S/AS01B | RTS, S/AS02A | Rabipur (Rabies) Vaccine
Number analyzed (Participants) | 61 | 62 | 66
titers | 593.7 [317.0 to 1111.9] | 635.8 [341.9 to 1182.5] | 28.6 [13.8 to 59.1]

20. Other Pre Specified Outcome: Geometric Mean Titers (GMTs) for Anti-HBs Antibodies by Infection Status PRE
Description: Geometric mean titers (GMTs) for Anti-HBs antibodies by infection status (Total Cohort) Infection defined as P. falciparum asexual parasitemia >0 PRE= Prevaccination
Time Frame: Prevaccination
Population: The Total Vaccinated Cohort includes all vaccinated subjects for whom data were available. For GMTs by infection status arms have been combined.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- Geometric Mean Antibody: Geometric Mean Antibody titer calculated on all subjects
Arm/Group | Geometric Mean Antibody
Number analyzed (Participants) | 163
titer
  Non-infected: PRE: number analyzed (Participants) | 67
  Non-infected: PRE | 11.1 [5.7 to 21.6]
  Infected: PRE: number analyzed (Participants) | 96
  Infected: PRE | 13.5 [7.9 to 22.9]

21. Other Pre Specified Outcome: Geometric Mean Titers (GMTs) for Anti-HBs Antibodies by Infection Status PIII (D90)
Description: Geometric mean titers (GMTs) for Anti-HBs antibodies by infection status (Total Cohort) Infection defined as P. falciparum asexual parasitemia >0 PIII(D90)= post dose 3 (day 90)
Time Frame: Day 90
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Geometric Mean Antibody
Number analyzed (Participants) | 152
titer
  Non-infected: PIII(D90): number analyzed (Participants) | 57
  Non-infected: PIII(D90) | 1558.3 [744.7 to 3260.7]
  Infected: PIII(D90): number analyzed (Participants) | 95
  Infected: PIII(D90) | 1532.6 [844.2 to 2782.4]

22. Other Pre Specified Outcome: Geometric Mean Titers (GMTs) for Anti-HBs Antibodies by Infection Status PIII (M12)
Description: Geometric mean titers (GMTs) for Anti-HBs antibodies by infection status (Total Cohort) Infection defined as P. falciparum asexual parasitemia >0 PIII(M12)= post dose 3 (month 12)
Time Frame: Month 12
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Geometric Mean Antibody
Number analyzed (Participants) | 132
titer
  Non-infected: PIII(M12): number analyzed (Participants) | 47
  Non-infected: PIII(M12) | 765.8 [384.8 to 1524.3]
  Infected: PIII(M12): number analyzed (Participants) | 85
  Infected: PIII(M12) | 499.0 [293.1 to 849.5]

23. Other Pre Specified Outcome: Geometric Mean Titers (GMTs) for Anti-CS Antibodies up to Month 12 by Vaccine Group PRE
Description: Geometric mean titers (GMTs) for Anti-CS antibodies accessed prevaccination, 1 month post dose 2, 1 month post dose 3, 4 months post dose 3 and 10 months post dose 3 PRE= prevaccination
Time Frame: Prevaccination
Population: Immunogenicity (According to protocol (ATP) Cohort): 222 subjects (75 RTS,S/AS01B, 74 RTS,S/AS02A, 73 rabies vaccine)
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | RTS, S/AS01B | RTS, S/AS02A | Rabipur (Rabies) Vaccine
Number analyzed (Participants) | 75 | 74 | 73
titers | 2.2 [1.6 to 2.9] | 1.2 [0.9 to 1.6] | 1.9 [1.4 to 2.5]

24. Other Pre Specified Outcome: Geometric Mean Titers (GMTs) for Anti-CS Antibodies up to Month 12 by Vaccine Group PII (D60)
Description: Geometric mean titers (GMTs) for Anti-CS antibodies accessed prevaccination, 1 month post dose 2, 1 month post dose 3, 4 months post dose 3 and 10 months post dose 3 PII(D60)= post dose 2 (day 60)
Time Frame: 1 month post dose 2
Population: Immunogenicity (According to protocol (ATP) Cohort): 222 subjects (75 RTS,S/AS01B, 74 RTS,S/AS02A, 73 rabies vaccine)
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | RTS, S/AS01B | RTS, S/AS02A | Rabipur (Rabies) Vaccine
Number analyzed (Participants) | 75 | 74 | 73
titers | 31.6 [23.9 to 41.6] | 16.7 [12.9 to 21.7] | 1.8 [1.4 to 2.3]

25. Other Pre Specified Outcome: Geometric Mean Titers (GMTs) for Anti-CS Antibodies up to Month 12 by Vaccine Group PIII (D90)
Description: Geometric mean titers (GMTs) for Anti-CS antibodies accessed prevaccination, 1 month post dose 2, 1 month post dose 3, 4 months post dose 3 and 10 months post dose 3 PIII(D90)= post dose 3 (day 90)
Time Frame: 1 month post dose 3
Population: Immunogenicity (According to protocol (ATP) Cohort): 213 subjects (72 RTS,S/AS01B, 72 RTS,S/AS02A, 69 rabies vaccine)
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | RTS, S/AS01B | RTS, S/AS02A | Rabipur (Rabies) Vaccine
Number analyzed (Participants) | 72 | 72 | 69
titers | 41.4 [31.7 to 54.2] | 21.4 [16.0 to 28.7] | 1.1 [1.1 to 2.0]

26. Other Pre Specified Outcome: Geometric Mean Titers (GMTs) for Anti-CS Antibodies up to Month 12 by Vaccine Group PIII (M6.5)
Description: Geometric mean titers (GMTs) for Anti-CS antibodies accessed prevaccination, 1 month post dose 2, 1 month post dose 3, 4 months post dose 3 and 10 months post dose 3 PIII(M6.5)= post dose 3 (month 6.5)
Time Frame: 4 months post dose 3
Population: Immunogenicity (According to protocol (ATP) Cohort): 207 subjects (69 RTS,S/AS01B, 69 RTS,S/AS02A, 69 rabies vaccine)
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | RTS, S/AS01B | RTS, S/AS02A | Rabipur (Rabies) Vaccine
Number analyzed (Participants) | 69 | 69 | 69
titers | 23.1 [17.1 to 31.1] | 13.1 [9.7 to 17.7] | 1.5 [1.1 to 2.0]

27. Other Pre Specified Outcome: Geometric Mean Titers (GMTs) for Anti-CS Antibodies up to Month 12 by Vaccine Group PIII (M12)
Description: Geometric mean titers (GMTs) for Anti-CS antibodies accessed prevaccination, 1 month post dose 2, 1 month post dose 3, 4 months post dose 3 and 10 months post dose 3 PIII(M12)= post dose 3 (month 12)
Time Frame: 10 months post dose 3
Population: Immunogenicity (According to protocol (ATP) Cohort): 189 subjects (61 RTS,S/AS01B, 62 RTS,S/AS02A, 66 rabies vaccine)
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | RTS, S/AS01B | RTS, S/AS02A | Rabipur (Rabies) Vaccine
Number analyzed (Participants) | 61 | 62 | 66
titers | 14.2 [10.7 to 18.9] | 7.3 [5.2 to 10.2] | 1.7 [1.3 to 2.3]

28. Other Pre Specified Outcome: Geometric Mean Antibody Titers (GMTs) for Anti-CS Antibodies by Infection Status PRE
Description: Geometric mean antibody titers (GMTs) for Anti-CS antibodies by infection status on RTS,S/AS01B and RTS,S/AS02A recipients only Infection defined as P. falciparum asexual parasitemia >0 PRE= Pre-vaccination
Time Frame: PRE
Population: The ATP Cohort includes all evaluable subjects for whom data were available. For GMTs by infection status arms have been combined.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Groups:
- Geometric Mean Antibody Titer: GMTs calculated on all subjects
Arm/Group | Geometric Mean Antibody Titer
Number analyzed (Participants) | 153
titers
  Infected: PRE: number analyzed (Participants) | 56
  Infected: PRE | 1.2 [0.9 to 1.7]
  Non-infected: PRE: number analyzed (Participants) | 97
  Non-infected: PRE | 2.0 [1.6 to 2.6]

29. Other Pre Specified Outcome: Geometric Mean Antibody Titers (GMTs) for Anti-CS Antibodies by Infection Status PII (D60)
Description: Geometric mean antibody titers (GMTs) for Anti-CS antibodies by infection status on RTS,S/AS01B and RTS,S/AS02A recipients only Infection defined as P. falciparum asexual parasitemia >0 PII(D60)= post dose 2 (day 60)
Time Frame: post dose 2 (day 60)
Population: as for outcome 28
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Geometric Mean Antibody Titer
Number analyzed (Participants) | 153
titers
  Infected: PII(D60): number analyzed (Participants) | 56
  Infected: PII(D60) | 11.9 [8.4 to 17.0]
  Non-infected: PII(D60): number analyzed (Participants) | 97
  Non-infected: PII(D60) | 33.9 [28.1 to 40.9]

30. Other Pre Specified Outcome: Geometric Mean Antibody Titers (GMTs) for Anti-CS Antibodies by Infection Status PIII (D90)
Description: Geometric mean antibody titers (GMTs) for Anti-CS antibodies by infection status on RTS,S/AS01B and RTS,S/AS02A recipients only Infection defined as P. falciparum asexual parasitemia >0 PIII(D90)= post dose 3 (day 90)
Time Frame: post dose 3 (day 90)
Population: as for outcome 28
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Geometric Mean Antibody Titer
Number analyzed (Participants) | 151
titers
  Infected: PIII(D90): number analyzed (Participants) | 56
  Infected: PIII(D90) | 18.3 [12.7 to 26.5]
  Non-infected: PIII(D90): number analyzed (Participants) | 95
  Non-infected: PIII(D90) | 40.1 [32.6 to 49.2]

31. Other Pre Specified Outcome: Geometric Mean Antibody Titers (GMTs) for Anti-CS Antibodies by Infection Status PIII (M6.5)
Description: Geometric mean antibody titers (GMTs) for Anti-CS antibodies by infection status on RTS,S/AS01B and RTS,S/AS02A recipients only Infection defined as P. falciparum asexual parasitemia >0 PIII(M6.5)= post dose 3 (month 6.5)
Time Frame: post dose 3 (month 6.5)
Population: as for outcome 28
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Geometric Mean Antibody Titer
Number analyzed (Participants) | 143
titers
  Infected: PIII(M6.5): number analyzed (Participants) | 54
  Infected: PIII(M6.5) | 9.9 [6.7 to 14.6]
  Non-infected: PIII(M6.5): number analyzed (Participants) | 89
  Non-infected: PIII(M6.5) | 25.1 [20.3 to 31.0]

32. Other Pre Specified Outcome: Seropositivity Rates for Anti-CS Antibodies by Vaccine Group PRE
Description: Seropositivity rates for Anti-CS antibodies accessed prevaccination, 1 month post dose 2, 1 month post dose 3, 4 months post dose 3 and 10 months post dose 3
  PRE= prevaccination
Time Frame: Prevaccination
Population: Immunogenicity (ATP Cohort): 222 subjects (75 RTS,S/AS01B, 74 RTS,S/AS02A, 73 rabies vaccine)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RTS, S/AS01B | RTS, S/AS02A | Rabipur (Rabies) Vaccine
Number analyzed (Participants) | 75 | 74 | 73
percentage of participants | 86.7 [76.8 to 93.4] | 75.7 [64.3 to 84.9] | 84.9 [74.6 to 92.2]

33. Other Pre Specified Outcome: Seropositivity Rates for Anti-CS Antibodies by Vaccine Group PII (D60)
Description: Seropositivity rates for Anti-CS antibodies accessed prevaccination, 1 month post dose 2, 1 month post dose 3, 4 months post dose 3 and 10 months post dose 3.
  PII(D60)= post dose 2 (day 60)
Time Frame: 1 month post dose 2
Population: Immunogenicity (According to protocol (ATP) Cohort): 222 subjects (75 RTS,S/AS01B, 74 RTS,S/AS02A, 73 rabies vaccine)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RTS, S/AS01B | RTS, S/AS02A | Rabipur (Rabies) Vaccine
Number analyzed (Participants) | 75 | 74 | 73
percentage of participants | 98.7 [92.8 to 100] | 100 [95.1 to 100] | 84.9 [74.6 to 92.2]

34. Other Pre Specified Outcome: Seropositivity Rates for Anti-CS Antibodies by Vaccine Group PIII (D90)
Description: Seropositivity rates for Anti-CS antibodies accessed prevaccination, 1 month post dose 2, 1 month post dose 3, 4 months post dose 3 and 10 months post dose 3
  PIII(D90)= post dose 3 (day 90)
Time Frame: 1 month post dose 3
Population: Immunogenicity (According to protocol (ATP) Cohort): 213 subjects (72 RTS,S/AS01B, 72 RTS,S/AS02A, 69 rabies vaccine)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RTS, S/AS01B | RTS, S/AS02A | Rabipur (Rabies) Vaccine
Number analyzed (Participants) | 72 | 72 | 69
percentage of participants | 98.6 [92.5 to 100] | 100 [95.0 to 100] | 82.6 [71.6 to 90.7]

35. Other Pre Specified Outcome: Seropositivity Rates for Anti-CS Antibodies by Vaccine Group PIII (M6.5)
Description: Seropositivity rates for Anti-CS antibodies accessed prevaccination, 1 month post dose 2, 1 month post dose 3, 4 months post dose 3 and 10 months post dose 3
  PIII(M6.5)= post dose 3 (month 6.5)
Time Frame: 4 months post dose 3
Population: Immunogenicity (According to protocol (ATP) Cohort): 207 subjects (69 RTS,S/AS01B, 69 RTS,S/AS02A, 69 rabies vaccine)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RTS, S/AS01B | RTS, S/AS02A | Rabipur (Rabies) Vaccine
Number analyzed (Participants) | 69 | 69 | 69
percentage of participants | 98.6 [92.2 to 100] | 98.6 [92.2 to 100] | 79.7 [68.3 to 88.4]

36. Other Pre Specified Outcome: Seropositivity Rates for Anti-CS Antibodies by Vaccine Group PIII (M12)
Description: Seropositivity rates for Anti-CS antibodies accessed prevaccination, 1 month post dose 2, 1 month post dose 3, 4 months post dose 3 and 10 months post dose 3
  PIII(M12)= post dose 3 (month 12)
Time Frame: 10 months post dose 3
Population: Immunogenicity (According to protocol (ATP) Cohort): 189 subjects (61 RTS,S/AS01B, 62 RTS,S/AS02A, 66 rabies vaccine)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RTS, S/AS01B | RTS, S/AS02A | Rabipur (Rabies) Vaccine
Number analyzed (Participants) | 61 | 62 | 66
percentage of participants | 100 [94.1 to 100] | 95.2 [86.5 to 99.0] | 80.3 [68.7 to 89.1]

37. Other Pre Specified Outcome: Seropositivity Rates for Anti-CS Antibodies by Infection Status PRE
Description: Seropositivity rates for Anti-CS antibodies by infection status on RTS,S/AS01B and RTS,S/AS02A recipients only Seropositive: >0.5EU/mL Infection defined as P. falciparum asexual parasitemia >0 PRE= Pre-vaccination
Time Frame: Prevaccination
Population: The ATP Cohort includes all evaluable subjects for whom data were available. For seropositivity rates by infection status arms have been combined.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Seropositive: Seropositive: >0.5 EU/mL
Arm/Group | Seropositive
Number analyzed (Participants) | 153
percentage of participants
  % of Infected: PRE: number analyzed (Participants) | 56
  % of Infected: PRE | 76.8 [63.6 to 87.0]
  % of Non-infected: PRE: number analyzed (Participants) | 97
  % of Non-infected: PRE | 83.5 [74.6 to 90.3]

38. Other Pre Specified Outcome: Seropositivity Rates for Anti-CS Antibodies by Infection Status PII (D60)
Description: Seropositivity rates for Anti-CS antibodies by infection status on RTS,S/AS01B and RTS,S/AS02A recipients only Seropositive: >0.5EU/mL Infection defined as P. falciparum asexual parasitemia >0 PII(D60)= post dose 2 (day 60)
Time Frame: post dose 2 (day 60)
Population: as for outcome 37
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Seropositive
Number analyzed (Participants) | 153
percentage of participants
  % of Infected: PII(D60): number analyzed (Participants) | 56
  % of Infected: PII(D60) | 98.2 [90.4 to 100]
  % of Non-infected: PII(D60): number analyzed (Participants) | 97
  % of Non-infected: PII(D60) | 100 [96.3 to 100]

39. Other Pre Specified Outcome: Seropositivity Rates for Anti-CS Antibodies by Infection Status PIII (D90)
Description: Seropositivity rates for Anti-CS antibodies by infection status on RTS,S/AS01B and RTS,S/AS02A recipients only Seropositive: >0.5EU/mL Infection defined as P. falciparum asexual parasitemia >0 PIII(D90)= post dose 3 (day 90)
Time Frame: post dose 3 (day 90)
Population: as for outcome 37
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Seropositive
Number analyzed (Participants) | 151
percentage of participants
  % of Infected: PIII(D90): number analyzed (Participants) | 56
  % of Infected: PIII(D90) | 98.2 [90.4 to 100]
  % of Non-infected: PIII(D90): number analyzed (Participants) | 95
  % of Non-infected: PIII(D90) | 100 [96.2 to 100]

40. Other Pre Specified Outcome: Seropositivity Rates for Anti-CS Antibodies by Infection Status PIII (M6.5)
Description: Seropositivity rates for Anti-CS antibodies by infection status on RTS,S/AS01B and RTS,S/AS02A recipients only Seropositive: >0.5EU/mL Infection defined as P. falciparum asexual parasitemia >0 PIII(M6.5)= post dose 3 (month 6.5)
Time Frame: post dose 3 (month 6.5)
Population: as for outcome 37
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Seropositive
Number analyzed (Participants) | 143
percentage of participants
  % of Infected: PIII(M6.5): number analyzed (Participants) | 54
  % of Infected: PIII(M6.5) | 98.1 [90.1 to 100]
  % of Non-infected: PIII(M6.5): number analyzed (Participants) | 89
  % of Non-infected: PIII(M6.5) | 98.9 [93.9 to 100]

41. Other Pre Specified Outcome: Efficacy: Vaccine Efficacy Against P. Falciparum Infection
Description: Number of subjects with an episode of parasitemia (first recording of infection of asexual stage falciparum parasites >0 detected by active detection of infection (ADI) or passive case detection)
Time Frame: 14 days after dose 3 and extending for 14 weeks
Population: Efficacy (According to protocol (ATP) Cohort): 228 subjects (74 RTS,S/AS01B, 79 RTS,S/AS02A, 75 rabies vaccine).
Measure: Number; unit: participants
Arm/Group | RTS, S/AS01B | RTS, S/AS02A | Rabipur (Rabies) Vaccine
Number analyzed (Participants) | 74 | 79 | 75
participants | 28 | 28 | 37

42. Other Pre Specified Outcome: Percentage of Participants With Positive and Negative Parasite Density
Description: Percentage of participants with positive and negative parasite density at month 6.5
Time Frame: at month 6.5
Population: Efficacy (According to protocol (ATP) Cohort): 228 subjects (74 RTS,S/AS01B, 79 RTS,S/AS02A, 75 rabies vaccine). Missing subject data: S/AS01B = 4, S/AS02A = 6, Rabipur = 4
Measure: Number; unit: % of subjects
Arm/Group | RTS, S/AS01B | RTS, S/AS02A | Rabipur (Rabies) Vaccine
Number analyzed (Participants) | 74 | 79 | 75
% of subjects
  Parasite Density: % of Negative Subjects | 91.4 | 93.2 | 95.8
  Parasite Density: % of Positive Subjects | 8.6 | 6.8 | 4.2

43. Other Pre Specified Outcome: Geometric Mean Antibody Titers (GMTs) of Asexual P. Falciparum Parasitemia
Description: Geometric Mean Antibody Titers (GMTs) of Asexual P. falciparum parasitemia at Month 6.5
Time Frame: Month 6.5
Population: Efficacy (According to protocol (ATP) Cohort): 228 subjects (74 RTS,S/AS01B, 79 RTS,S/AS02A, 75 rabies vaccine).
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | RTS, S/AS01B | RTS, S/AS02A | Rabipur (Rabies) Vaccine
Number analyzed (Participants) | 74 | 79 | 75
titers | 1122 [-525.0 to 2769.0] | 342 [-115.4 to 799.8] | 711 [-846.8 to 2268.8]

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- (RTS, S/AS01B): RTS, S/AS01B: 0.5mL dose; 50ug RTS, S antigen, 50ug QS21 and liposomes in phosphate-buffered saline administered intramuscular deltoid of non-dominant arm at 0, 1 and 2 months.
  RTS, S/AS01B: 0.5mL dose; 50ug RTS, S antigen, 50ug QS21 and liposomes in phosphate-buffered saline administered intramuscular deltoid of non-dominant arm at 0, 1 and 2 months.
- (RTS, S/AS02A): RTS, S/AS02A: 0.5mL dose; 50ug RTS, S antigen, 50ug QS21 and proprietary oil-water emulsion in phosphate-buffered saline administered intramuscular deltoid of non-dominant arm at 0, 1 and 2 months.
  RTS, S/AS02A: 0.5mL dose; 50ug RTS, S antigen, 50ug QS21 and proprietary oil-water emulsion in phosphate-buffered saline administered intramuscular deltoid of non-dominant arm at 0, 1 and 2 months.
- Rabipur (Rabies) Vaccine: Rabipur (Rabies) Vaccine: 1.0mL dose administered intramuscular deltoid of non-dominant arm at 0, 1 and 2 months
  Rabipur (Rabies) Vaccine: .0mL dose administered intramuscular deltoid of non-dominant arm at 0, 1 and 2 months
Arm/Group | (RTS, S/AS01B) | (RTS, S/AS02A) | Rabipur (Rabies) Vaccine
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/85 | 0/85
Serious Adverse Events (participants affected / at risk) | 5/85 | 1/85 | 5/85
Other Adverse Events (participants affected / at risk) | 81/85 | 82/85 | 82/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | (RTS, S/AS01B) (N=85) | (RTS, S/AS02A) (N=85) | Rabipur (Rabies) Vaccine (N=85)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Wound necrosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
HIV infection (Infections and infestations) | 2 (2) | 0 (0) | 3 (3)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Malaria (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Trichomoniasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Peptic Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Disseminated tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Meningitis cryptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalitis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | (RTS, S/AS01B) (N=85) | (RTS, S/AS02A) (N=85) | Rabipur (Rabies) Vaccine (N=85)
Fatigue (General disorders) | 35 (35) | 28 (28) | 26 (26)
Fever (General disorders) | 17 (17) | 11 (11) | 10 (10)
Gastrointestinal (Gastrointestinal disorders) | 37 (37) | 33 (33) | 33 (33)
Headache (Nervous system disorders) | 54 (54) | 57 (57) | 45 (45)
Joint pain at other location (Musculoskeletal and connective tissue disorders) | 23 (23) | 19 (19) | 17 (17)
Muscle aches (Musculoskeletal and connective tissue disorders) | 21 (21) | 21 (21) | 24 (24)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 2 (2) | 3 (3) | 6 (6)
Ear pain (Ear and labyrinth disorders) | 6 (6) | 3 (3) | 2 (2)
Conjunctivitis (Eye disorders) | 10 (10) | 9 (9) | 8 (8)
Conjunctivitis allergic (Eye disorders) | 6 (6) | 9 (9) | 4 (4)
Eye pain (Eye disorders) | 0 (0) | 3 (3) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 7 (7) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 17 (17) | 17 (17) | 14 (14)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 4 (4) | 3 (3)
Anal skin tags (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Anal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Bowel sounds (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 6 (6)
Diarrhea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 3 (3) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 4 (4) | 0 (0) | 2 (2)
Glossitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperchlorhydria (Gastrointestinal disorders) | 4 (4) | 2 (2) | 2 (2)
Lip exfoliation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (4)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 3 (3) | 7 (7) | 3 (3)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 14 (14) | 9 (9) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Asthenia (General disorders) | 3 (3) | 0 (0) | 2 (2)
Chest pain (General disorders) | 9 (9) | 7 (7) | 12 (12)
Chills (General disorders) | 6 (6) | 4 (4) | 3 (3)
Fatigue (General disorders) | 2 (2) | 2 (2) | 4 (4)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 1 (1)
Hangover (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hunger (General disorders) | 0 (0) | 0 (0) | 1 (1)
Inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 7 (7) | 3 (3) | 4 (4)
Nodule (General disorders) | 1 (1) | 0 (0) | 2 (2)
Pain (General disorders) | 8 (8) | 4 (4) | 3 (3)
Pitting oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 15 (15) | 12 (12) | 11 (11)
Swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
Multiple allergies (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Amoebiasis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Ascariasis (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
Body tinea (Infections and infestations) | 6 (6) | 6 (6) | 5 (5)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Candidiasis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 3 (3) | 4 (4) | 4 (4)
Conjunctivitis infective (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Dental caries (Infections and infestations) | 7 (7) | 5 (5) | 4 (4)
Dysentery (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2) | 6 (6)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Genitourinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Giardiasis (Infections and infestations) | 7 (7) | 11 (11) | 9 (9)
Gonorrhea (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Helminthic infection (Infections and infestations) | 8 (8) | 7 (7) | 3 (3)
Herpes simplex (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Hookworm infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Impetigo (Infections and infestations) | 6 (6) | 7 (7) | 8 (8)
Laryngitis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 19 (19) | 14 (14) | 21 (21)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 2 (2) | 3 (3) | 1 (1)
Pharyngitis (Infections and infestations) | 7 (7) | 5 (5) | 9 (9)
Pneumonia (Infections and infestations) | 5 (5) | 3 (3) | 1 (1)
Pulpitis dental (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Rhinitis (Infections and infestations) | 12 (12) | 8 (8) | 9 (9)
Schistosomiasis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Septic rash (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sexually transmitted disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Strongyloidiasis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Tinea capitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Tinea cruris (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tinea infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tinea versicolour (Infections and infestations) | 3 (3) | 1 (1) | 4 (4)
Tonsillitis (Infections and infestations) | 4 (4) | 4 (4) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Trichomoniasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Typhoid fever (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 50 (50) | 54 (54) | 48 (48)
Urethritis (Infections and infestations) | 3 (3) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2) | 3 (3)
Vaginal candidiasis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Vulvovaginitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Wound sepsis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 6 (6)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 14 (14) | 18 (18) | 20 (20)
Wound (Injury, poisoning and procedural complications) | 5 (5) | 3 (3) | 5 (5)
Mean cell volume decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 25 (25) | 15 (15) | 19 (19)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (11) | 5 (5) | 10 (10)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (16) | 13 (13) | 20 (20)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (11) | 9 (9) | 13 (13)
Neck pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 4 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 3 (3)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 9 (9) | 3 (3) | 5 (5)
Headache (Nervous system disorders) | 24 (24) | 32 (32) | 37 (37)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Balanitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 2 (2)
Genital ulceration (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Mammory duct ectasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cough epistaxis (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 11 (11) | 10 (10)
Epixtaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (7) | 10 (10)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 10 (10) | 4 (4)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Rash pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No